CLINICAL TRIAL: NCT03203369
Title: Phase 1, Open-label Dose-escalation and Dose-expansion Study to Evaluate the Safety, Expansion, Persistence and Clinical Activity of a Single Dose of UCART123 (Allogeneic Engineered T-cells Expressing Anti-CD123 Chimeric Antigen Receptor), Administered in Patients With Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN)
Brief Title: Study to Evaluate the Safety and Clinical Activity of UCART123 in Patients With BPDCN
Acronym: ABC123
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was discontinued due to sponsor's decision and not a consequence of any safety concern.
Sponsor: Cellectis S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCART123_02
Record Dates: First submitted 2017-06-14; First posted 2017-06-29 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN)
Keywords: Blastic plasmacytoid dendritic cell neoplasm; Natural Killer (NK) cell blastic lymphoma; Hematologic malignancies; Cluster of differentiation (CD) CD4+CD56+ hematodermic tumor; Acute leukemia and myeloid neoplasms; Chimeric Antigen Receptor T-cell (CAR-T) therapy; Allogeneic; Cluster of differentiation 4 (CD4); Cluster of differentiation 56 (CD56)
MeSH Terms: conditions — Blastic Plasmacytoid Dendritic Cell Neoplasm; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): A single intravenous administration of UCART123. Dose escalation in Part 1 will include 3 doses ranging from 6.25 x 10^5 cells/kg to 6.25 x 10^6 cells/kg and continue until the Recommended Phase 2 Dose (RP2D) is identified.
  Interventions: Biological: UCART123
- Part 2: Dose Expansion (Experimental): A single intravenous administration of UCART123 at the RP2D. 2 Cohorts: Patients with Relapsed/Refractory BPDCN and Newly Diagnosed BPDCN.
  Interventions: Biological: UCART123

INTERVENTIONS:
Biological: UCART123 — Allogeneic engineered T-cells expressing anti-CD123 Chimeric Antigen Receptor given as a single dose following a lymphodepleting regimen.

SUMMARY:
A Phase 1 dose-finding study of Universal Chimeric Antigen Receptor T-cells targeting cluster of differentiation (CD) 123 (UCART123) administered intravenously to patients with relapsed or refractory Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN), followed by a dose expansion phase in relapsed or refractory BPDCN patients or newly diagnosed BPDCN patients.

ELIGIBILITY:
Main Inclusion Criteria:

* Patients with a diagnosis BPDCN according to World Health Organization (WHO) classification confirmed by hematopathology;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Incidence, nature, and severity of adverse events and serious adverse events | Through day 84

CONTACTS AND LOCATIONS:
Overall Officials: Ioana Kloos, MD, Study Director — Cellectis S.A.
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided